CLINICAL TRIAL: NCT04648553
Title: A Pilot Randomized Control Trial of the Task-Based Grounding Program
Brief Title: Task-Based Grounding Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, James T. Craig, Assistant Professor of Psychiatry, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D21019
Record Dates: First submitted 2020-11-14; First posted 2020-12-01 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Aggressive; Defiant Disorder, Oppositional; Attention Deficit Hyperactivity Disorder
Keywords: Oppositional Defiant Disorder; Behavioral Parent Training
MeSH Terms: conditions — Aggression; Oppositional Defiant Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Task-Based Grounding (Experimental): Participating parents will be provided with three 50-minute Task Based Grounding sessions using a standardized manual over 6 weeks.
  Interventions: Behavioral: Task-Based Grounding
- Connected Care (Enhanced treatment as usual) (Sham Comparator): Participating parents will be provided with two sessions and one phone check-in call over 6 weeks. They will work with a "care navigator" to assess their child's needs, find them an appropriate referral for care, and help problem solve barriers to finding a therapist.
  Interventions: Behavioral: Connected Care (Enhanced Treatment as usual)

INTERVENTIONS:
Behavioral: Task-Based Grounding — Three 50 minutes sessions with an interventionist that includes 6 non-punitive components of treatment common in Behavioral Parent Trainings: Education on behavior change, positive one-on-one time between parents and their children, differential attending to positive and negative behaviors, effective praise, giving effective instructions, and using a point and reward system to encourage prosocial behaviors. These components are distilled into 5 skill modules and paired with Task-Based Grounding, which involves a brief restriction of privileges and provides children with the opportunity to end the restriction by completing a prosocial task.
  Arms: Task-Based Grounding
Behavioral: Connected Care (Enhanced Treatment as usual) — Two sessions with a facilitator. The facilitator does NOT provide any guidance to the parent on managing their child's behavior, but provides empathy and problem solving to help them find a resource that best fits their needs. It is particularly geared towards helping parents connect with Behavioral Parent Trainings to address the needs of children with oppositional, defiant, or aggressive behaviors.
  Arms: Connected Care (Enhanced treatment as usual)

SUMMARY:
The purpose of this study is to improve the availability of brief interventions to help children with defiant, aggressive and disruptive behaviors by creating a brief scalable intervention for parents delivered via telehealth. As phase 1 study, we are conducting a 2-arm pilot feasibility RCT in order the intervention, measures, and procedures to be used in a larger efficacy trial. The first arm will include a 3-session behavioral therapy treatment we call Task-Based Grounding and the second arm will be an enhanced treatment as usual comparison group.

DETAILED DESCRIPTION:
The investigators have developed a 3-session psychosocial intervention for parents of children between 9-14 with disruptive behaviors. The intervention uses telehealth visits along with written and online resources to teach them parent management skills. To evaluate the acceptability of this intervention and the feasibility of our methods, the investigators will recruit 20 parent-child dyads to participate in this study. This is a mixed methods pilot feasibility RCT design. The investigators designed this study to test the acceptability of the intervention to parents and test the feasibility of our recruitment, retention, measurement, and delivery mechanisms for both the experimental and comparison conditions. The investigators will use a block randomization method to separate parent-child dyads into either treatment or comparison groups. The treatment condition involves 3 telehealth visits and a set of parenting resources. The enhanced treatment as usual condition will involve contact with a "care navigator" that will assess behavior problems in the child and help the parents find an appropriate referral to care in their community. Both groups will be followed for 10 weeks, provide outcome data, and participate in semi-structured qualitative interviews to accept acceptability.

ELIGIBILITY:
Inclusion Criteria:

* Participating parent-child dyads must include a child between the ages of 9-14 years old and adult over the age of 18.
* The child must have a Vanderbilt Oppositional Defiant Disorder score >3
* The participating caregiver must be a legal guardian of participating child

Exclusion Criteria (child refers to the primary participant's child)

* Child ever been hospitalized for a psychiatric problem
* Child ever attempted suicide or stated that they had a plan to attempt suicide within the past year.
* Child ever engaged in self-harm behaviors
* Child has significant legal history such as adjudicated of a crime or been in diversion
* Child has ever been diagnosed with: Obsessive Compulsive Disorder, Post Traumatic Stress Disorder, Intellectual Disability or Developmental Delay, Speech or Hearing Delay, Autism Spectrum Disorder, Schizophrenia or another psychotic disorder, A substance abuse disorder (or had serious concerns about substance use).
* Parent can communicate in spoken English
* Parent is under the age of 18.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of referred participants | Through study completion, approximately 5 months.
  Feasibility of recruitment will be measured by number of participants referred
Number of participants who screen positive | Through study completion, approximately 5 months.
  Feasibility of recruitment will be measured by number of participants who screen positive
Change from Baseline Session attendance at visit 3 | Session attendance will be taken at Session 1 (week 0) and Session 3 (week 6)
  Feasibility of the participant retention in the program will be measured by session attendance by participants
Number of participants enrolled | Through study completion, approximately 5 months.
  Feasibility of recruitment will be measured by number of participants enrolled
Number of participants who complete all assessment measures | Through study completion, approximately 5 months.
  Feasibility of assessment measures will be measured by number of participants who complete assessment measures
Fidelity of the training provided | Through study completion, approximately 5 months.
  as measured by having a trained listener code and score fidelity using a checklist developed specifically for the content of each session. Audio recording of intervention sessions will be used. There are 35 items on the checklist, each worth 1pt. Score will be in terms of percentage, with a minimum score of 0 and a maximum score 100%.
Intervention acceptability as measured by the Treatment Evaluation Inventory Short Form | Follow-up/post intervention (up to 10 weeks)
  as measured by Treatment Evaluation Inventory Short Form post intervention which measures intervention acceptance. The established cut off scores for determining if a treatment is acceptable is a score of 27. Min score possible is 0, max score possible is 32. Higher scores indicate greater acceptability.
Intervention Acceptability as measured by the Therapy Attitude Inventory | Follow-up/post intervention (up to 10 weeks)
  as measured by the Therapy Attitude Inventory post intervention which measures acceptability of behavioral parent trainings. Min score of 1 is possible, max score of 50 is possible. Higher scores indicate greater acceptability.
Intervention Acceptability as measured by the Participant Experiences Questionnaire | Follow-up/post intervention (up to 10 weeks)
  as measured by the Participant Experiences Questionnaire which measures acceptability of each skill module included in the program and is specific to program content. Min score of 0 possible, max score of 36 possible. Higher scores indicate greater acceptability.
Acceptability as measured by qualitative interview | Follow-up/post intervention (up to 10 weeks)
  as measured by 30 minute semi-structured qualitative interview with participants conducted by a research assistant trained and supervised by the study PI

SECONDARY OUTCOMES:
Adherence to the intervention | Available for completion every day for 10 weeks
  as measured by daily logs that track both children's aggressive and defiant behaviors and parenting behaviors. A count of each time a parent used a skill from the program will be used to estimate adherence and assess whether they matched the appropriate skills to the reported misbehaviors.

CONTACTS AND LOCATIONS:
Overall Officials: James T Craig, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No